CLINICAL TRIAL: NCT06462079
Title: A Phase II Clinical Study of Sacituzumab Govitecan Combined With Head Radiotherapy for the Treatment of Brain Metastases From Her2-negative Breast Cancer
Brief Title: Sacituzumab Govitecan Combined With Head Radiotherapy for Her2-negative Breast Cancer Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-028-01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Brain Metastasis
Keywords: Breast cancer; Her2- (Human Epidermal Growth Factor Receptor 2 Negative); Brain metastasis; Sacituzumab Govitecan; Radiation therapy
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms | interventions — sacituzumab govitecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Experimental): Patients were treated with Sacituzumab Govitecan 10 mg/kg in 21-day treatment cycles with intravenous infusions on days 1 and 8 and continued until disease progression or unacceptable toxicity. Radiotherapy was administered after the second infusion of Sacituzumab Govitecan, on day 9 after the start of this regimen. The radiotherapy regimen was: brain metastases at a dose of 60 Gy/20 doses. For lesions located adjacent to the brainstem and optic nerve, 54 Gy/20 doses were given. For patients with ≥5 lesions, whole-brain radiotherapy at 40 Gy/20 doses was synchronized with radiotherapy to localized brain metastases.
  Interventions: Drug: Sacituzumab Govitecan; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Patients were treated with Sacituzumab Govitecan 10 mg/kg in 21-day treatment cycles with intravenous infusions on days 1 and 8 and continued until disease progression or unacceptable toxicity.
  Other Names: Trodelvy
Radiation: Radiotherapy — Radiotherapy was administered after the second infusion of Sacituzumab Govitecan, on day 9 after the start of this regimen. The radiotherapy regimen was: brain metastases at a dose of 60 Gy/20 doses. For lesions located adjacent to the brainstem and optic nerve, 54 Gy/20 doses were given. For patients with ≥5 lesions, whole-brain radiotherapy at 40 Gy/20 doses was synchronized with radiotherapy to localized brain metastases.

SUMMARY:
The incidence of brain metastasis of Her2-negative breast cancer is high, which seriously affects the prognosis of patients.The treatment of brain metastasis of Her2-negative breast cancer is still tricky. The local efficacy of head radiotherapy for breast cancer brain metastases is remarkable, and systemic tumor progression in patients with brain metastases is the main reason for treatment failure. Sacituzumab Govitecan is the only Trop-2 antibody-coupled drug (ADC) approved for the treatment of unresectable locally advanced or metastatic Her2-negative breast cancer. However, the objective remission rate of Sacituzumab Govitecan for intracranial metastatic lesions has not been satisfactory. This study is an open, uncontrolled phase II clinical study to observe the efficacy and safety of Sacituzumab Govitecan combined with intracranial radiotherapy in the treatment of patients with brain metastases from Her2-negative breast cancer, in order to find a more effective treatment method.

DETAILED DESCRIPTION:
This study is a single-arm open phase II clinical trial. It aims to observe the effectiveness and safety of Sacituzumab Govitecan combined with head radiotherapy in the treatment of Her2-negative breast cancer brain metastases, and to search for a more effective treatment option for Her2-negative breast cancer brain metastases. Patients were treated with Sacituzumab Govitecan 10mg/kg every 21 days as a treatment cycle, which was infused intravenously on day 1 and day 8, and the treatment was continued until the disease progressed or unacceptable toxicity occurred. Radiotherapy was administered after the second infusion of Sacituzumab Govitecan, on day 9 after the start of this regimen. The radiotherapy regimen was: brain metastases at a dose of 60 Gy/20 doses. For lesions located adjacent to the brainstem and optic nerve, 54 Gy/20 doses were given. For patients with ≥5 lesions, whole-brain radiotherapy at 40 Gy/20 doses was synchronized with radiotherapy to localized brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Have a definitive pathologic diagnosis of breast cancer with subtype Her2- (including IHC 0, IHC 1+ or IHC 2+ and ISH negative);
2. Have a measurable intracranial lesion;
3. Age ≥ 18 years;

Exclusion Criteria:

1. Patients with cerebrospinal membrane metastases;
2. Patients with acute/subacute hemorrhagic metastasis;
3. Inadequate organ function: 1) Blood tests: ANC ≤ 1.5 x 10^9/L, PLT ≤ 90 x 10^9/L, Hb ≤ 90g/L; 2) Blood biochemistry tests: TBIL ≥ 1.5 times the upper limit of normal; 3) ALT and AST ≥ 2.5 times the upper limit of normal;
4. Presence of serious and/or uncontrolled comorbidities that may affect participation: 1) allergy to study medications or adjuvant materials; 2) history of immunodeficiency, including HIV-positive or other acquired or congenital immunodeficiency diseases; 3) serious concomitant illnesses;
5. Pregnant and lactating female patients; female patients of childbearing age who are unwilling to use effective contraception during the trial period;
6. Patients who are unable to complete enhanced contrast MRI;
7. Patients who have been treated with Sacituzumab Govitecan and are resistant to the drug;
8. Any other condition that, in the opinion of the investigator, makes the patient ineligible for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
1-year CNS progression-free survival (NPFS) | From the time patients receive this treatment until the next 1 year
  Proportion of patients free of CNS progression at 1 year from the time the patient receives this treatment. Neurological progression was assessed according to the Response Assessment of Neuro-Oncology Brain Metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
Intracranial objective remission rate (IORR) | Assessed at 2 months after the end of treatment or at the time of patient death
  The proportion of patients whose brain metastases shrink in volume to achieve complete remission/partial remission from the time the patient receives this treatment. Complete remission/partial remission is assessed according to the Response Assessment of Neuro-Oncology Brain Metastases (RANO-BM) criteria
Rate of new intracranial lesions | Assessed 2 months after the end of treatment or at the time of patient's death
  The proportion of patients presenting with new brain metastases from the time the patient received treatment. New brain metastases are assessed according to the Response Assessment of Neuro-Oncology Brain Metastases (RANO-BM) criteria.
Overall progression-free survival (PFS) | All patients received at least 6 months of follow-up, and NPFS was assessed from the start of treatment to the date of the first documented progression of an extracranial lesion or the date of death from any cause, whichever came first.
  The time from the time the patient receives this treatment to the time of disease progression or death. Assessment of extracranial lesions follows the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1).
Overall survival | Assessments were performed at least 7 months after diagnosis of brain metastases or before death
  Survival time was recorded from the date of patient enrollment. All patients were followed until death or the end of the study.
Incidence of Treatment-Related Adverse Events | Assessments were performed 2 months after the end of treatment or at the time of the patient's death
  The incidence of treatment-related adverse events was measured to determine tolerability and safety. Adverse events (AEs) were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03).Grade 3-5 events were defined as moderate and severe adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, Principal Investigator — Huizhou Hospital of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: Individual participant data will be public accessable via contacting with principal investigator by email within 6 months after the trial complete.

REFERENCES:
- [Background] Tarantino P, Carmagnani Pestana R, Corti C, Modi S, Bardia A, Tolaney SM, Cortes J, Soria JC, Curigliano G. Antibody-drug conjugates: Smart chemotherapy delivery across tumor histologies. CA Cancer J Clin. 2022 Mar;72(2):165-182. doi: 10.3322/caac.21705. Epub 2021 Nov 12. PMID 34767258
- [Background] Ocean AJ, Starodub AN, Bardia A, Vahdat LT, Isakoff SJ, Guarino M, Messersmith WA, Picozzi VJ, Mayer IA, Wegener WA, Maliakal P, Govindan SV, Sharkey RM, Goldenberg DM. Sacituzumab govitecan (IMMU-132), an anti-Trop-2-SN-38 antibody-drug conjugate for the treatment of diverse epithelial cancers: Safety and pharmacokinetics. Cancer. 2017 Oct 1;123(19):3843-3854. doi: 10.1002/cncr.30789. Epub 2017 May 30. PMID 28558150
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Loirat D, Tredan O, Ciruelos E, Dalenc F, Gomez Pardo P, Jhaveri KL, Delaney R, Valdez T, Wang H, Motwani M, Yoon OK, Verret W, Tolaney SM. Overall survival with sacituzumab govitecan in hormone receptor-positive and human epidermal growth factor receptor 2-negative metastatic breast cancer (TROPiCS-02): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Oct 21;402(10411):1423-1433. doi: 10.1016/S0140-6736(23)01245-X. Epub 2023 Aug 23. PMID 37633306
- [Background] Bardia A, Hurvitz SA, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Sardesai SD, Kalinsky K, Zelnak AB, Weaver R, Traina T, Dalenc F, Aftimos P, Lynce F, Diab S, Cortes J, O'Shaughnessy J, Dieras V, Ferrario C, Schmid P, Carey LA, Gianni L, Piccart MJ, Loibl S, Goldenberg DM, Hong Q, Olivo MS, Itri LM, Rugo HS; ASCENT Clinical Trial Investigators. Sacituzumab Govitecan in Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2021 Apr 22;384(16):1529-1541. doi: 10.1056/NEJMoa2028485. PMID 33882206
- [Background] Xu B, Ma F, Wang T, Wang S, Tong Z, Li W, Wu X, Wang X, Sun T, Pan Y, Yao H, Wang X, Luo T, Yang J, Zeng X, Zhao W, Cong XJ, Chen J. A Phase IIb, single arm, multicenter trial of sacituzumab govitecan in Chinese patients with metastatic triple-negative breast cancer who received at least two prior treatments. Int J Cancer. 2023 May 15;152(10):2134-2144. doi: 10.1002/ijc.34424. Epub 2023 Jan 30. PMID 36621000